CLINICAL TRIAL: NCT02082938
Title: The Use of a Brace to Retrain Hemiparetic Gait in Patients With Genu Recurvatum: Effects on Plantar Pressure Distribution
Brief Title: The Use of Brace to Retrain Hemiparetic Gait
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Éder Kröeff Cardoso, PT Éder Kröeff Cardoso Master Degree, Federal University of Health Science of Porto Alegre
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Eder01
Record Dates: First submitted 2014-03-04; First posted 2014-03-10 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2012-03

CONDITIONS: Stroke Nos Without Residual Deficits
Keywords: stroke,; rehabilitation,; hemiparesis,; gait training
MeSH Terms: conditions — Stroke; Paresis | interventions — Braces

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bracing (Experimental): Bracing: the patients began four weeks of training the gait with the brace, under the guidance and observation of the physiotherapist belonging to the group of authors of this study.
  Interventions: Device: Bracing

INTERVENTIONS:
Device: Bracing — Twice a week, for a period of 5 weeks, before the sessions in the physiotherapy clinic the patients participating in the study were asked to walk at a self-selected speed on flat ground along a corridor 50 meters long, with the brace being used for fifteen minutes of gait retraining of the affected side.

SUMMARY:
The purpose of this study is to verify if the incorporation of a new brace, which assists in gait rehabilitation, can contribute to the rehabilitation process for stroke patients.

DETAILED DESCRIPTION:
Objective To compare the behavior of plantar pressure peak distribution, before and after training using a brace for gait rehabilitation.

Method The brace was developed with the aim of promoting better biomechanical alignment, as well as providing proprioceptive information in order to stimulate action in the knee's flexor muscle groups, thus facilitating the activation pattern contrary to what occurs during genu recurvatum. We conducted a quasi-experimental "before and after" study with twelve hemiparetic adult patients who had genu recurvatum in the gait. The plantar pressure peaks were compared at the various moments of the study.

ELIGIBILITY:
Inclusion Criteria:

* the presence of hemiparesis after the stroke, with an evolution time of between 6 and 24 months, the ability to walk without using assistive aids, and the presence of genu recurvatum during the mid-stance in the gait.

Exclusion Criteria:

* conditions that would preclude evaluation and training with the brace; for example, the presence of contractures or fixed deformities in the lower limbs, and moderate to severe impairments related to cognition, perception, attention, or language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-03; Primary Completion 2012-04 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
distribution of plantar pressures during walking | 4 weeks
  To evaluate the distribution of plantar pressures during walking, for individuals with hemiparesis, before and after training with a brace for gait retraining and control of genu recurvatum.
  To observe the gait evolution of 12 patientes after the trainnig with a orthotic device.

CONTACTS AND LOCATIONS:
Overall Officials: Éder K Cardoso, Master, Principal Investigator — Federal University of Health Science of Porto Alegre